CLINICAL TRIAL: NCT04240015
Title: Association of Periodontitis With Oral Health Related Quality of Life
Status: Completed | Type: Observational
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Mehtap Bilgin Çetin, Dr. Mehtap Bilgin Çetin, Baskent University
Other Study IDs: Mehtap
Record Dates: First submitted 2020-01-17; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Periodontitis, Adult
Keywords: oral health related quality of life; periodontal disease
MeSH Terms: conditions — Chronic Periodontitis; Periodontal Diseases | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Periodontitis: Periodontitis group consisted of patients diagnosed with periodontitis
  Interventions: Other: Oral-Dental Health-Related Quality of Life-United Kingdom (OHRQoL-UK) scale
- Patients without periodontitis: Patients without periodontitis group constituted patients without periodontitis
  Interventions: Other: Oral-Dental Health-Related Quality of Life-United Kingdom (OHRQoL-UK) scale

INTERVENTIONS:
Other: Oral-Dental Health-Related Quality of Life-United Kingdom (OHRQoL-UK) scale — It consists of 4 different categories and 16 questions evaluating the effects of OHRQoL in positive and negative areas. These categories are as follows; symptoms (2 questions), physical status (5 questions), psychological status (5 questions), social status (4 questions) ' Questions on the OHRQoL-UK scale were scored using the Likert-type scale as 'very bad effect-score 1, bad effect-score 2, no effect-score 3, good effect-score 4, very good effect-score 5. The scores obtained from all questions were summed to give the scores of the 4 sub-categories separately and the total OHRQoL score. A higher total score indicates a higher OHRQoL.

SUMMARY:
Objective: The aim of this study was to investigate the impact of periodontitis on oral health-related quality of life (OHQoL) and the factors may associated with OHQoL.

Methods: 50 untreated periodontitis patients and 50 individuals without periodontitis were enrolled in the study. All subjects underwent detailed periodontal examination and probing depth (PD), clinical attachment level (CAL) measurements were performed. OHRQoL was assessed through the Oral Health Quality of Life-United Kingdom (OHRQoL-UK) scale. Symptoms of periodontitis was determined by Visual Analogue Scale (VAS). Socio-demographic characteristics, medical history, smoking status, hygiene habits of the all individuals were recorded.

DETAILED DESCRIPTION:
The primary aim of the present study was to compare the scores of OHQoL-UK of patients with periodontitis to who didn't have periodontitis/healthy controls. Our second aim was investigate the factors (education, smoking, gender, periodontal clinical parameters) may related to oral health related quality of life).

Materials and methods Study group The present clinical study was conducted with a study group of 50 untreated periodontitis patients and a control group of 50 individuals without periodontitis (age and gender matched) who applied to Hacettepe University Faculty of Dentistry Department of Periodontology. Clinical examination and evaluation of patients' complaint All participants underwent comprehensive periodontal examination by a calibrated and masked examiner. probing pocket depth (PPD = distance between gingival margin and bottom of the periodontal pocket) and clinical attachment level (CAL = distance between the cement-enamel junction and bottom of the periodontal pocket) were evaluated. All periodontal measurements were recorded at six sites around each tooth by a periodontal probe excluding third molar.The patients' complaints/symptoms associated with periodontitis (gingival bleeding and edema, halitosis, flaring, mobile teeth, gingival hyperemia, bad taste, dentin/root sensitivity) were also evaluated by using Visual Analogue Scale [VAS (0-10)]. In the evaluation with VAS, a straight line of 100 mm was used on the vertical axis and the starting and ending points were numbered 0 and 100. Individuals were asked to what extent they perceived the symptoms of periodontitis and were asked to make an evaluation between 0 and 100 on the scale and to put an x mark on the scale. In the evaluation of the scale, the marking point of the patient was measured with a caliper from the beginning of the scale.

Assesment of OHRQoL OHRQoL was assessed using the Oral-Dental Health-Related Quality of Life-United Kingdom (OHRQoL-UK) scale. It consists of 4 different categories and 16 questions evaluating the effects of OHRQoL in positive and negative areas. These categories are as follows; symptoms (2 questions), physical status (5 questions), psychological status (5 questions), social status (4 questions) ' Questions on the OHRQoL-UK scale were scored using the Likert-type scale as 'very bad effect-score 1, bad effect-score 2, no effect-score 3, good effect-score 4, very good effect-score 5. The scores obtained from all questions were summed to give the scores of the 4 sub-categories separately and the total OHRQoL score. A higher total score indicates a higher OHRQoL.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 18 years and older
* Patients have at least 20 remaining teeth

Exclusion Criteria:

* Individuals who have received periodontal treatment in the last 6 months individuals (anti-inflammatory, antibiotic, etc.)
* Pregnancy
* Subjects with systemic disease and who used any medication that may affect the periodontal condition in the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The present clinical study was conducted with a study group of 50 untreated periodontitis patients and a control group of 50 individuals without periodontitis (age and gender matched) who applied to Hacettepe University Faculty of Dentistry Department of Periodontology.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-10-05; Primary Completion 2014-01-10 (Actual); Study Completion 2014-02-12 (Actual)

PRIMARY OUTCOMES:
OHRQoL-UK scores of the study population | 20 minutes
  OHRQoL was assessed using the Oral-Dental Health-Related Quality of Life-United Kingdom (OHRQoL-UK) scale.It consists of 4 different categories and 16 questions that evaluate the effects of OHRQoL in both positive and negative areas. These categories are listed as follows; symptoms (2 questions), physical status (5 questions), psychological status (5 questions), social status (4 questions) ' Questions on the OHRQoL-UK scale were scored using the Likert-type scale as 'very bad effect-score 1, bad effect-score 2, no effect-score 3, good effect-score 4, very good effect-score 5. The scores were gathered from all surveys and they were summarized to give the scores of 4 sub-categories separately, along with the total OHRQoL score. A higher total score indicates a higher OHRQoL.

SECONDARY OUTCOMES:
Complaints of study population. | 5 minutes
  Patient complaints and symptoms associated with periodontitis, which is characterized by gingival bleeding and edema, halitosis, flaring, mobile teeth, gingival hyperemia, bad taste and dentin/root sensitivity, were also evaluated using Visual Analogue Scale [VAS (0-10)]. In VAS evaluation, a straight line of 100 mm was used on the vertical axis and the starting and ending points were numbered as 0 and 100. Individuals were asked to assess to what extent they perceived the symptoms of periodontitis. They were requested to make an evaluation between 0 and 100 scale and mark that scale. Patient's score was measured with a caliper from the beginning of the scale.